CLINICAL TRIAL: NCT02988531
Title: Validation of PET-MRI for Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AC16105
Record Dates: First submitted 2016-09-23; First posted 2016-12-09 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2017-10

CONDITIONS: MRI; PET Scan; Positron-Emission Tomography; Cardiovascular Disease; Coronary Artery Disease; Magnetic Resonance Imaging
Keywords: PET; MRI; Attenuation; Correction; Cardiovascular; coronary; disease
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PET/MR (Experimental): Participants to have PET/MR scan
  Interventions: Other: PET/MR scan

INTERVENTIONS:
Other: PET/MR scan — Patients to undergo PET/MR scanning after PET/CT scan. Patients will have had an injection of 18F Sodium Fluoride for their PET/CT therefore will not need another dose of radiotracer prior to their PET/MR scan.

SUMMARY:
To determine whether PET-MRI can obtain comparable images to PET-CT in those with coronary artery disease.

DETAILED DESCRIPTION:
Positron emission tomography (PET) is method of non-invasively imaging a metabolic process. It has been used in clinical medicine for many years with its primary use in identifying areas of increased metabolic activity as possible cancers. It involves the use of a radionuclide (or radiotracer) labelled to a chemical involved in a certain metabolic process. In order for the PET signal from the radiotracer to be detected by the scanner the radionuclide emits a small dose of ionizing radiation. Examples of commonly used radionuclides include 18FDG and 18 Sodium Fluoride (18NaF). In order to locate where exactly these areas of abnormal or increased metabolic activity were, Computerised Tomography (CT) has traditionally been used for anatomical correlation.

Until recently PET-CT has largely been confined for use in oncology. More recently however PET-CT has been utilized to detect vulnerable plaques in those with coronary artery disease. In coronary artery disease 18F-fluoride acts as a marker of novel calcification activity within the plaque. Similar to other conditions, calcification in coronary atheroma occurs as a healing response to intense necrotic inflammation, making 18F- fluoride a useful marker of high-risk atherosclerotic plaque. This has been demonstrated in those with stable angina as well as localizing the culprit plaque in those with myocardial infarction in 90% of cases.

Magnetic resonance imaging is being increasingly adopted in cardiovascular imaging and holds particular attraction due to its ability to provide information about soft tissue structures both with and without contrast agents, as well as its safety due to absence of exposure to ionising radiation and rapid imaging speed, which is useful in a moving organ like the heart.

PET-MR works differently to PET-CT. PET relies on the annihilation of protons with electrons, generating 511 keV photons, which are absorbed in bodily tissues differently depending on their electron density (e.g. heart denser than lungs). Because of this PET images can appear brighter or darker in different tissues. To account for this, a technique of attenuation correction is employed. This is usually in the form of what is called a transmission scan (low intensity CT scan) which grades tissue density and corrects the PET signal accordingly. Given MRI measures proton density and not electron density different attenuation correction techniques are needed. It has not yet been established how best to do this despite multiple efforts using differing techniques.

Previous single centre studies have demonstrated the feasibility of MRI-PET. The technique's translation to clinical practice has been limited due to the global lack of reliable attenuation correction methods. During his recent Clinical Research Imaging Fellowship in New York, co-investigator (Dr Dweck) developed a novel free breathing method of attenuation correction in a combined PET-MR scanner that reduced scanning time and improved efficiency and has shown immense promise. In Edinburgh a similar combined PET-MR scanner (mMR, Siemens, Erlangen, Germany) has been installed, but have not yet replicated or validated this technique. If the investigators can demonstrate and apply a method of attenuation correction that is acceptable and shows good comparability of MRI-PET to PET-CT images they may be able to use this imaging method as an alternative to PET-CT.

Benefits which may translate clinically include superior soft tissue characterisation and significantly reduced radiation dosages. The technique could be applied across a range of medical conditions in addition to cardiovascular disease and oncology.

The investigators are hopeful to establish a suitable attenuation correction method so that PET-MR can match or even supersede PET-CT as an imaging technique providing accurate biological, anatomical and functional information in those with cardiovascular disease with low radiation doses.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing thoracic PET-CT scans (this can include NHS and patients enrolled in other research studies)
* Aged over 50 years old. No upper age limit
* Provision of informed consent prior to any study specific procedures

Exclusion Criteria:

* Inability or unwilling to give informed consent.
* Major intercurrent illness with life-expectancy <2 years.
* Contra-indication to Magnetic resonance imaging.
* Permanent or persistent atrial fibrillation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-09 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
The standard uptake values (SUV's) of volumes of interest (VOI's) on corresponding PET-CT and PET-MR images will be evaluated by expert. The distribution of PET positive VOI's will be compared using a cut-off of 1.6 for tissue to background ratio (TBR). | 7 months

SECONDARY OUTCOMES:
Standard breath-held MR-based attenuation correction will be compared to a novel free-breathing approach. Impact on PET image artifacts and the interpretation of vascular uptake will be evaluated semi-quantitatively by expert readers. | 7 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Edinburgh, Edinburgh, Lothian, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plans to share patient specific data

REFERENCES:
- [Background] Dweck MR, Chow MW, Joshi NV, Williams MC, Jones C, Fletcher AM, Richardson H, White A, McKillop G, van Beek EJ, Boon NA, Rudd JH, Newby DE. Coronary arterial 18F-sodium fluoride uptake: a novel marker of plaque biology. J Am Coll Cardiol. 2012 Apr 24;59(17):1539-48. doi: 10.1016/j.jacc.2011.12.037. PMID 22516444
- [Background] Dweck MR, Khaw HJ, Sng GK, Luo EL, Baird A, Williams MC, Makiello P, Mirsadraee S, Joshi NV, van Beek EJ, Boon NA, Rudd JH, Newby DE. Aortic stenosis, atherosclerosis, and skeletal bone: is there a common link with calcification and inflammation? Eur Heart J. 2013 Jun;34(21):1567-74. doi: 10.1093/eurheartj/eht034. Epub 2013 Feb 7. PMID 23391586
- [Background] Joshi NV, Vesey AT, Williams MC, Shah AS, Calvert PA, Craighead FH, Yeoh SE, Wallace W, Salter D, Fletcher AM, van Beek EJ, Flapan AD, Uren NG, Behan MW, Cruden NL, Mills NL, Fox KA, Rudd JH, Dweck MR, Newby DE. 18F-fluoride positron emission tomography for identification of ruptured and high-risk coronary atherosclerotic plaques: a prospective clinical trial. Lancet. 2014 Feb 22;383(9918):705-13. doi: 10.1016/S0140-6736(13)61754-7. Epub 2013 Nov 11. PMID 24224999